CLINICAL TRIAL: NCT04979338
Title: Development of Effective, Opioid Sparing Techniques for Peri-operative Pain Management of Transgender Patients Undergoing Gender Affirming Surgeries
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Maurice M. Garcia, Director of the Cedars-Sinai Transgender Surgery and Health Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000879
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gender Dysphoria
Keywords: Gender Dysphoria; Gender-Affirming Surgery; Peri-Operative Pain; Pain Management; Surgery Pain; Sex Reassignment Surgery; Gender Reassignment Surgery; Vaginoplasty; Phalloplasty; Quality Improvement; Opioid Use
MeSH Terms: conditions — Gender Dysphoria; Agnosia | interventions — Bupivacaine; Dental Occlusion; Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1 (Active Comparator): Depending on which one of the thirteen possible gender-affirming surgeries the participant is undergoing, a combination of the following anesthetic block(s) will be used in this arm at either the pre-incision, intra-op, mid-surgery, end of surgery, or continuous time points:
  * Bilateral spermatic cord block (0.5% bupivacaine, 10cc per spermatic cord)
  * Local anesthetic (0.25% or 0.5% bupivacaine + 1:200K epinephrine)
  * Bilateral ultrasound guided pudendal nerve block (20-40 cc of 0.25% bupivacaine + 1:200K epinephrine)
  * Ultrasound guided Continuous Infraclavicular Brachial Plexus Block
  * Ultrasound guided Continuous Femoral Nerve Block
  * Pecs I & II Block (0.25% bupivacaine: 15-30ml per side for Pecs I-III)
  Interventions: Other: Ultrasound guided Continuous Infraclavicular Brachial Plexus Block; Other: Ultrasound guided Continuous Femoral Nerve Block; Other: Ultrasound guided Pudendal Nerve Block; Drug: Bupivacaine; Other: Bilateral spermatic cord block; Other: Pecs I & II Block; Other: Local anesthetic
- Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #2 (Active Comparator): Depending on which one of the thirteen possible gender-affirming surgeries the participant is undergoing, a combination of the following anesthetic block(s) will be used in this arm at either the intra-op, post-op, or end of surgery time points:
  * Bilateral ultrasound-guided Transversus Abdominis Plane Block (40-60cc of 0.25% bupivacaine with 1:200K epinephrine)
  * Local anesthetic (0.25 or 0.5% bupivacaine + 1:200K epinephrine)
  Interventions: Drug: Bupivacaine; Other: Bilateral ultrasound guided Transversus Abdominis Plane Block; Other: Local anesthetic
- Surgery-specific general anesthetic + local anesthetic at incision site (Active Comparator): Depending on which one of the thirteen possible gender-affirming surgeries the participant is undergoing, a combination of the following anesthetic block(s) will be used in this arm at either the mid-surgery or end of surgery time points:
  * Bilateral spermatic cord block (0.5% bupivacaine, 10cc per spermatic cord)
  * Local anesthetic (0.25 or 0.5% bupivacaine + 1:200K epinephrine)
  Interventions: Drug: Bupivacaine; Other: Bilateral spermatic cord block; Other: Local anesthetic

INTERVENTIONS:
Other: Ultrasound guided Continuous Infraclavicular Brachial Plexus Block — 20cc of 0.25% bupivacaine + 1:200K epinephrine will be administered at start of case, 20cc of 0.25% bupivacaine + 1:200K epinephrine at end of case, and 6cc/hr of 0.25% bupivacaine at post-op [administered by anesthesiologist]
  Arms: Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1
Other: Ultrasound guided Continuous Femoral Nerve Block — 20cc of 0.25% bupivacaine + 1:200K epinephrine will be administered at start of case, 20cc of 0.25% bupivacaine + 1:200K epinephrine at end of case, and 6cc/hr of 0.25% bupivacaine at post-op [administered by anesthesiologist]
  Arms: Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1
Other: Ultrasound guided Pudendal Nerve Block — 20-40cc of 0.25% bupivacaine + 1:200K epinephrine [administered by anesthesiologist, pre-incision]
  Arms: Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1
Drug: Bupivacaine — 0.25% or 0.5% with or without 1:200K epinephrine
  Other Names: Marcaine
Other: Bilateral ultrasound guided Transversus Abdominis Plane Block — 40-60cc of 0.25% bupivacaine + 1:200K epinephrine [administered by anesthesiologist post-op or at end of surgery]
  Arms: Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #2
Other: Bilateral spermatic cord block — 10cc per spermatic cord of 0.5% bupivacaine [administered by surgeon @ intraop]
  Arms: Surgery-specific general anesthetic + local anesthetic at incision site; Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1
Other: Pecs I & II Block — 0.25% bupivacaine: 15-30mL per side for Pecs I-III
  Arms: Surgery-specific general anesthetic + ultrasound guided peripheral nerve block #1
Other: Local anesthetic — 0.25% or 0.5% bupivacaine into the appropriate surgical site

SUMMARY:
This study will compare the current standard-of-care pain treatment regimen options that are available to patients who undergo gender-affirming surgery. The purpose of this research is to determine if any of these options are more (versus less) effective than the others to manage surgery related pain, after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Transgender persons 18 years and older
* Undergoing gender affirming surgeries performed by either Dr. Maurice Garcia (orchiectomy only, vaginoplasty with or without canal & orchiectomy, colon-vaginoplasty, & peritoneal vaginoplasty; Stage I phalloplasty, or stage II phalloplasty); Dr. Edward Ray (feminizing chest surgery, masculinizing chest surgery, stage I phalloplasty); Dr. Amit Gupta (orchiectomy and peritoneal vaginoplasty only); or Dr. Yosef Nasseri (colon vaginoplasty surgery)

Exclusion Criteria:

* Patients who do not meet the inclusion criteria above
* Any contraindications to the study drugs.
* Patients with neurologic deficits that preclude them from sensing pain.
* Patients with implanted pain neuromodulator devices (e.g., neurostimulator)
* Patients who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender persons
Enrollment: 640 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in peri-operative pain location and intensity over time, as measured by anatomic pain maps | Any time pain is experienced, starting on the morning of post-operative Day 1 to End of Study at the final post-operative visit (average of 30 days after surgery)
  Anterior and posterior illustrations of the body, with pre-defined areas involved in surgery that may be circled, will be used to define pain location. Pain scores for each circled area will be measured on a Likert-scale between 0-10, with 0 indicating no pain and 10 indicating the worst pain experienced in respondent's life.
Changes in opioid consumption per 24 hours, measured by total inpatient and total outpatient | Per 24 hours, starting on post-operative Day 1 to End of Study at the final post-operative visit (average of 30 days after surgery)
  Inpatient opioid consumption will be obtained from hospital records. Outpatient opioid consumption will be determined from completed medication logs. Opioid consumption will be measured per 24 hours, by hospital location (e.g., PACU versus Ward), and by post-operative day.
Change in the opioid side effect of urinary retention, as indicated by time to spontaneous voiding | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  Recorded time to spontaneous voiding will be collected from hospital records.
Change in the opioid side effect of urinary retention, as measured by a Urinary Bother Symptom Score Questionnaire | Pre-operative visit, Discharge (average of 7 days after surgery), and End of Study/final post-operative visit (average of 30 days after surgery)
  A Urinary Bother Symptom Score Questionnaire, obtained from the American Urological Association, will assess the frequency of different urinary problems, such as incomplete emptying, intermittency, and urgency. Each urinary problem will be measured on a scale from 0 to 5, with 0 indicating "none/not at all" and 5 indicating "almost always."
Change in the opioid side effect of decreased GI motility and ileus, as indicated by number of post-operative days until commencement of regular passage of flatus | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  Recorded number of post-operative days until commencement of regular passage of flatus will be obtained from hospital records.
Change in the opioid side effect of nausea, as indicated by number of post-operative days to toleration of liquid diet and regular diet, as well as reported experience of nausea | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  Recorded number of post-operative days and experience of nausea will be obtained from hospital records.
Post-operative length of inpatient stay | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  Length of inpatient stay will be obtained from hospital records as the recorded number of days spent inpatient after surgery
Global satisfaction with respect to pain and physical comfort, as measured by a Quality of Recovery 15-Item Inventory | Daily, starting on the morning of post-operative Day 1 to End of Study at the final post-operative visit (average of 30 days after surgery)
  Questions 1-10 will assess global well-being and physical comfort, such as ability to return to work or usual home activities, feeling rested, ability to enjoy food, and general feelings of well-being. These questions will be rated on a scale of 0 to 10, with 0 indicating none of the time (poor) and 10 indicating all of the time (excellent).
  Questions 11-15 will assess pain and physical comfort, such as presence of moderate/severe pain, nausea or vomiting, worried or anxious feelings, and sad or depressed feelings. These questions will be rated on a scale of 0 to 10, with 0 indicating all of the time (poor) and 10 indicating none of the time (excellent).
Frequency of treatment complications | End of study (average of 30 days after surgery)
  Treatment complications, such as hematoma, infection, etc., will only include those that are determined to be related to the study treatment.

SECONDARY OUTCOMES:
Time to mobilization | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  The recorded number of days to mobilization will be obtained from hospital records.
Time to first day of bowel movement | Post-operative Day 1 to Discharge (average of 7 days after surgery)
  The recorded number of days to first bowel movement will be obtained from hospital records.
Number of participants with any hospital readmission within 30 days of discharge | 30 days after Day of Discharge (average of 7 days after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Maurice M Garcia, M.D., MAS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center - North and South Towers, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No